CLINICAL TRIAL: NCT06964152
Title: Prospective Use of Computational Cardiac Imaging Analysis to Guide Ventricular Tachycardia Ablation Procedures (AI-VT)
Brief Title: Computational Cardiac Imaging Analysis to Guide Ventricular Tachycardia Ablation Procedures (AI-VT)
Acronym: AI-VT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Gordon Ho, Principal Investigator, Cardiac Electrophysiology Physician, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 171964
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Ventricular Tachycardia (VT); Premature Ventricular Contraction (PVC); Ventricular Fibrillation
Keywords: electrocardiography, arrhythmia mapping, 3D mapping, electroanatomic mapping, cardiac computed tomography, artificial intelligence, computational modeling
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- VT ablation guided by supplemental non-invasive computational imaging analysis (Experimental): The electrophysiologist performing the standard-of-care VT ablation will have access to supplemental arrhythmia targeting/localization information provided by computational non-invasive ECG and/or cardiac CT imaging analysis
  Interventions: Diagnostic Test: Computational electrocardiography and cardiac computed tomography mapping

INTERVENTIONS:
Diagnostic Test: Computational electrocardiography and cardiac computed tomography mapping — Use of non-invasive computational ECG and cardiac CT models to localize arrhythmia origins

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes (clinical efficacy and safety) of using supplemental non-invasive computational ECG and cardiac imaging analysis tools to help guide ablation of ventricular tachycardia.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 100
2. Evidence of ventricular tachycardia on ECG, telemetry or by CIED interrogation.

Exclusion Criteria:

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrent ventricular tachycardia | 1 year
  Ventricular tachycardia episodes defined as implantable cardioverter defibrillator (ICD) therapies (anti-tachycardia pacing and shocks)
All-cause death | 1 year

SECONDARY OUTCOMES:
Acute hemodynamic decompensation | 24 hours post-op
  acute development of hypotension, cardiogenic shock, escalation of inotropes/pressors, or need for unplanned percutaneous hemodynamic support
Unplanned prolonged ICU upgrade | 48 hours
  In outpatient elective cases, change in patient condiction neccessitating unplanned ICU upgrade lasting longer than 48 hours.
acute cerebrovascular accident (embolic) | 24 hours post-op
acute pericardial tamponade requiring intervention | 24 hours post-op
  new expanding hemorrhagic pericardial effusion causing tamponade requiring urgent pericardiocentesis
vascular complication requiring intervention | 24 hours post-op
  vascular access complication (bleeding or occlusion) requiring blood transfusion or vascular procedure (such as peripheral angioplasty)

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited de-identified clinical datasets may be shared upon individual request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1/1/2029-12/31/2032

REFERENCES:
- [Background] Krummen DE, Villongco CT, Ho G, Schricker AA, Field ME, Sung K, Kacena KA, Martinson MS, Hoffmayer KS, Hsu JC, Raissi F, Feld GK, McCulloch AD, Han FT. Forward-Solution Noninvasive Computational Arrhythmia Mapping: The VMAP Study. Circ Arrhythm Electrophysiol. 2022 Sep;15(9):e010857. doi: 10.1161/CIRCEP.122.010857. Epub 2022 Sep 7. PMID 36069189